CLINICAL TRIAL: NCT00628238
Title: A Two-Arm, Multi-center Trial of Revlimid® and Rituximab, for First-Line Treatment in Patients With B-cell Chronic Lymphocytic Leukemia (CLL)
Brief Title: Multi-center Trial of Revlimid® and Rituximab, for First-Line Treatment of Chronic Lymphocytic Leukemia (CLL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chronic Lymphocytic Leukemia Research Consortium (Network)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Thomas J. Kipps, M.D., Ph.D., Chronic Lymphocytic Leukemia Research Consortium (CRC)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRC014; Celgene # RV-CLL-PI-0223
Expanded Access: Available
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Lymphocytic Leukemia; CLL; Untreated; Front-line; First-Line; Initial Therapy
Keywords: Chronic Lymphocytic Leukemia Research Consortium; Chronic lymphocytic leukemia; CLL; CLL Research Consortium; CRC; Revlimid; lenalidomide; Rituximab; Rituxan; First-line; therapy; untreated; Frontline
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Subjects younger than 65 years old.
  Interventions: Drug: Lenalidomide and Rituximab
- B (Active Comparator): Subjects aged 65 years and older
  Interventions: Drug: Lenalidomide and Rituximab

INTERVENTIONS:
Drug: Lenalidomide and Rituximab — Lenalidomide starting at a low dose and escalated based on patient tolerability 21 days of every cycle. Rituximab at 375mg/m2 administered following the first 21 days of lenalidomide monotherapy, continued weekly throughout cycle 2, and then every 4 weeks for subsequent cycles. Each patient may receive up to a maximum of 7 cycles of treatment if no progressive disease or significant toxicity.
  Other Names: Revlimid; CC-5013; Rituxan
  Arms: A
Drug: Lenalidomide and Rituximab — Lenalidomide starting at a low dose and escalated based on patient tolerability 21 days of every cycle. Rituximab at 375mg/m2 administered following the first 21 days of lenalidomide monotherapy, continued weekly throughout cycle 2, and then every 4 weeks for subsequent cycles. Each patient may receive up to a maximum of 7 cycles of treatment if no progressive disease or significant toxicity.
  Other Names: Revlimid; CC-5013; Rituxan
  Arms: B

SUMMARY:
The study is a two-arm, multi-center trial of Revlimid® and Rituximab, for the frontline treatment of patients with Chronic Lymphocytic Leukemia (CLL) designed and conducted by the CLL Research Consortium (CRC). The purpose of this study is to determine the response rate of the combination of Revlimid® and Rituximab in previously untreated CLL patients in two arms- those aged 65 years and above and those younger than 65. Secondary objectives will evaluate the safety of the combination of Revlimid® and Rituximab, response duration, improvement in hematologic parameters, and the significance of the tumor flare reaction. All patients will have assessment of known prognostic factors for CLL as well as novel prognostic factors will be evaluated for predicting response to treatment. Biologic corollary studies are designed to evaluate the mechanism of Revlimid® in CLL and the combination of Revlimid® and Rituximab.

DETAILED DESCRIPTION:
The CLL Research Consortium (CRC) is conducting a two-arm, multi-center phase II trial of Revlimid® and rituximab for the first-line treatment of patients with CLL.

Revlimid® (lenalidomide) a derivative of thalidomide with immune-modulating properties. Revlimid® is FDA approved for treatment of relapsed multiple myeloma and 5q- myelodysplastic syndrome. Revlimid® has promising clinical activity in relapsed CLL in two early clinical trials. However, the mechanism(s) whereby Revlimid® is active in CLL is unknown. Rituximab (Rituxan®) is a protein that binds to CD20 expressed on normal and leukemia B cells. Rituximab is FDA approved for the treatment of lymphoma and is used commonly for the treatment of CLL. The purposes of this study are to evaluate the safety and activity of the combination of Revlimid® and rituximab in CLL, elucidate the mechanism of Revlimid® in CLL, and to assess whether prognostic factors might predict those patients likely to benefit from this therapy in the future.

As older patients are commonly under-represented in CLL clinical trials and are less tolerable of frontline therapy that utilizes combinations of fludarabine and cyclophosphamide the trial has two arms; one to specifically assess for the tolerability of the regimen in older subjects.

The primary objective of this study is to determine the response rate of the combination of Revlimid® and Rituximab in previously untreated CLL patients in two arms- those aged 65 years and above and those younger than 65. Secondary objectives will evaluate the safety of the combination of Revlimid® and Rituximab, response duration, improvement in hematologic parameters, activity of the combination in high-risk CLL subsets, and the significance of the tumor flare reaction.

All patients will have baseline assessment of known CLL prognostic factors including: immunoglobulin variable heavy chain (IgVH) gene mutational status, interphase cytogenetics, intracellular ZAP-70 expression, and CD38 expression through the CRC tissue core. These known prognostic features in CLL together with novel prognostic factors will be evaluated for the ability to predict response to treatment with Revlimid® and the combination of Revlimid® and Rituximab. Extensive biologic corollary studies are designed to evaluate the mechanism of Revlimid® in CLL, the impact of Revlimid® on the CLL microenvironment, and Revlimid®'s impact on and rituximab mediated cytotoxicity.

All patients will receive the same treatment. Revlimid® will be started at a low dose and slowly escalated based on patient tolerability. Rituximab will be administered following 21 days of Revlimid® monotherapy. Patients will continue treatment for up to 7 cycles unless there is toxicity or progressive disease. There are three planned response assessments for the subjects: a single agent Revlimid® response assessment prior to the addition of rituximab, after 3 cycles of treatment, and following all the therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of chronic lymphocytic leukemia with no history of previous treatments with monoclonal antibodies or chemotherapy.
2. Subjects must have an indication for treatment as defined by the NCI Working Group Guidelines
3. Understand and voluntarily sign an informed consent form.
4. Age ≥18 years at the time of signing the informed consent form.
5. Able to adhere to the study visit schedule and other protocol requirements.
6. ECOG performance status of ≤ 2 at study entry (see Appendix A).
7. Laboratory test results within these ranges: Absolute neutrophil count ≥ 1.0 x 109/L, Platelet count ≥ 50 x 109/L, Serum creatinine ≤ 1.5 mg/dL, Total bilirubin ≤ 1.5 mg/dL, AST & ALT ≤ 2 x ULN
8. Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
9. Disease free of prior malignancies for ≥ 2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "insitu" of the cervix or breast

Exclusion Criteria:

1. Previous treatment for CLL with chemotherapy or monoclonal antibodies
2. Known Hepatitis B Ag positive, Hepatitis C positive patients
3. Known HIV positive patients
4. Patients with uncontrolled Autoimmune Hemolytic Anemia (AIHA) or autoimmune thrombocytopenia (ITP).
5. Inability to provide informed consent.
6. Concurrent malignancy (excluding basal and squamous cell skin cancers).
7. Active fungal, bacterial, and/or viral infection.
8. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
9. Pregnant or breast-feeding females. (Lactating females must agree not to breast feed while taking lenalidomide).
10. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
11. Use of any other experimental drug or therapy within 28 days of baseline.
12. Known hypersensitivity to thalidomide.
13. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
14. Any prior use of lenalidomide.
15. Concurrent use of other anti-cancer agents or treatments.
16. Patients with history of deep venous thrombus or pulmonary embolism. Patients who are at increased risk of thrombosis during treatment with lenalidomide including those taking concurrent erythropoietin, darbepoetin or high-dose corticosteroids are also excluded.
17. Patients with a history of embolic events (e.g. TIA) from arrhythmia or peripheral arterial disease or of recent MI whether or not treated with anti-platelet drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Efficacy to be assessed by clinical response rate following 3 cycles of treatment and the NCI-CLL working group response rate assessed after completion of all treatment. | clinical response assessment after 3 cycles of therapy and 3 months following completion of all therapy for NCI-CLL working group response assessment

SECONDARY OUTCOMES:
Safety - type, frequency, severity, and relationship of adverse events to study treatment | Throughout the study period
Time To Progression | Following therapy until disease progression
Evaluate response to lenalidomide in relationship to molecular and genetic prognostic features in CLL; including ZAP-70 status, IgVH gene mutational status, and FISH. | Following final response assessment
Compare the efficacy and tolerability of the combination of Revlimid and rituximab for patients younger than 65 years, and for those 65 and older. • | following final response assessment
Evaluate change in hematological parameters including neutropenia, anemia, and thrombocytopenia following treatment with the combination of Revlimid and rituximab. | Following final response assessment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Kipps, M.D., Ph.D, Study Director — Director of the CLL Research Consortium and University of California San Diego; Danelle F James, M.D., Principal Investigator — CLL Research Consortium and University of California San Diego
Locations (5):
- United States (5):
  - University of California San Diego, La Jolla, California
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University, Columbus, Ohio
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas

REFERENCES:
- [Background] Chanan-Khan A, Miller KC, Musial L, Lawrence D, Padmanabhan S, Takeshita K, Porter CW, Goodrich DW, Bernstein ZP, Wallace P, Spaner D, Mohr A, Byrne C, Hernandez-Ilizaliturri F, Chrystal C, Starostik P, Czuczman MS. Clinical efficacy of lenalidomide in patients with relapsed or refractory chronic lymphocytic leukemia: results of a phase II study. J Clin Oncol. 2006 Dec 1;24(34):5343-9. doi: 10.1200/JCO.2005.05.0401. Epub 2006 Nov 6. PMID 17088571
- [Background] Chanan-Khan A, Porter CW. Immunomodulating drugs for chronic lymphocytic leukaemia. Lancet Oncol. 2006 Jun;7(6):480-8. doi: 10.1016/S1470-2045(06)70723-9. PMID 16750498
- [Background] Ferrajoli A, Lee BN, Schlette EJ, O'Brien SM, Gao H, Wen S, Wierda WG, Estrov Z, Faderl S, Cohen EN, Li C, Reuben JM, Keating MJ. Lenalidomide induces complete and partial remissions in patients with relapsed and refractory chronic lymphocytic leukemia. Blood. 2008 Jun 1;111(11):5291-7. doi: 10.1182/blood-2007-12-130120. Epub 2008 Mar 11. PMID 18334676
- See also: Website for the CLL Research Consortium — http://cllresearch.com/
- See also: Moore's UCSD Cancer Center — http://cancer.ucsd.edu/